CLINICAL TRIAL: NCT03054090
Title: Restoring Primary Care in Virginia: PCOR Learning as a Pathway to Value
Brief Title: Heart of Virginia Healthcare
Acronym: HVH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Virginia Center for Health Innovation (Unknown); Center for Health Policy Development (Unknown); George Mason University (Other); Health Quality Innovators (Unknown); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R18HS023913-01 (AHRQ)
Record Dates: First submitted 2016-09-22; First posted 2017-02-15 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular Diseases; Primary Care
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Quality Improvement support (Other): A blended support strategy will include practice facilitation, expert consultation, collaborative learning events, an online support center, and data feedback and benchmarking.
  Interventions: Other: Quality Improvement Support

INTERVENTIONS:
Other: Quality Improvement Support — Practices will receive a blended strategy of quality improvement facilitation to help participating practices incorporate PCOR clinical and organizational findings while building their overall practice capabilities. Primary care practices will be provided tools and training to improve the rates of screening and treatment of risk factors for heart attacks and strokes, as well as other chronic illnesses and the delivery of preventive services.

SUMMARY:
Most care for chronic conditions is provided by primary care clinicians. Although Virginia ranks 4th among the 50 states in average income, it ranks 27th in mortality due to heart attacks and strokes. The scope and focus of this project will materially improve the rates of screening and treatment of risk factors for heart attacks and strokes, and will give primary care clinicians the tools and training to improve the care of other chronic illnesses and the delivery of preventive services.

DETAILED DESCRIPTION:
Restoring Primary Care in Virginia: Patient Centered Outcomes Research (PCOR) Learning as a Pathway to Value is an extension of the Virginia Center for Health Innovation's (VCHI) work to address primary care transformation in its Virginia Health Innovation Plan. VCHI, in partnership with four of Virginia's schools of medicine, the Virginia Center for Health Quality (VHQC), and evaluation specialists at George Mason University, will form the Virginia Primary Care Transformation Collaborative (VPCTC). They will use an evidence-based, comprehensive strategy to help up to 300 small-to-medium sized primary care practices: 1) accelerate incorporation of PCOR clinical and organizational findings into practice with an initial focus on cardiovascular health and the Aspirin, Blood Pressure, Cholesterol, and Smoking (ABCS); 2) increase their capacity to integrate new PCOR findings on an on-going basis; and 3) learn strategies that can help them sustain and revitalize their organizations while restoring the joy to primary care practice. Practice supports will include on-site coaching, expert consultation, collaborative learning events, an online support center, and data feedback and benchmarking. As a result of this project, "Restoring Primary Care in Virginia," participating practices will develop stronger Quality Improvement (QI) capacity and learn strategies that can help them sustain and revitalize their organizations while restoring the joy to primary care practice. The value proposition to recruit and retain participating practices includes: Improved financial performance; improved clinician, staff, and patient satisfaction; objectively improved quality of care; improved ability to negotiate for and receive pay for performance bonuses, including Electronic Medical Record (EMR) meaningful use stage 2; completion of Part IV certification by the American Board of Family Medicine (ABFM) and American Board of Internal Medicine (ABIM) for QI work completed in this initiative; and engagement in a self-sustaining learning collaborative of similar practices after the end of the project. The evaluation plan is designed to answer these questions: (1) Did the VPCTC intervention improve the performance of small physician practices in Virginia as measured by the individual ABCS? (2) Which elements of the intervention were most important to the physicians for performance improvement? (3) Did "maintenance" or follow-up intervention activities add value or was the initial intense intervention enough to produce the measured impact? (4) Which internal contextual or structural features of practices at baseline are most likely to be associated with improved performance (e.g., expansive use of EMRs, degree of adaptive reserve or change processing capacity, number of physicians in the practice, etc.)? (5) Did the VPCTC improve the capacity of small physician practices to implement future PCOR findings and improve quality on an ongoing basis? (6) Which elements of the intervention were most important to the physicians for QI capacity building? Multivariate statistical modeling of clinical performance and survey data will be performed to answer questions 1, 3, and 4.

Qualitative interviews, surveys and statistical analysis of survey results will answer questions 2, 5, and 6.

ELIGIBILITY:
Inclusion Criteria:

* small to medium sized primary care practices in virginia that serve adults

Exclusion Criteria:

* large sized primary care practices
* pediatric practices

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2015-05; Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Aspirin prescriptions | 3 month
  Practice level rates of aspirin or other anti-thrombotics being prescribed. The outcome measure will be assessed from data extracted from practice EMR.
Blood pressure | 3 months
  Blood pressure control for hypertensives. The outcome measure will be assessed from data extracted from practice EMR.
Statin prescriptions | 3 months
  Practice level rates of Statins being prescribed for categories of higher risk cholesterol levels. The outcome measure will be assessed from data extracted from practice EMR.
Smoking | 3 months
  Smoking assessment. The outcome measure will be assessed from data extracted from practice EMR.
Smoking | 3 months
  Smoking cessation counseling. The outcome measure will be assessed from data extracted from practice EMR.

SECONDARY OUTCOMES:
Capacities to incorporate new patient centered outcome research | 1 year after intervention
  Capacities of practices to incorporate new patient centered outcome research into their care of patients. This outcome measure will be assessed using surveys.
Capacities to incorporate new patient centered outcome research | 1 year after intervention
  Capacities of practices to incorporate new patient centered outcome research into their care of patients. This outcome measure will be assessed using interviews.
Joy in practice | 1 year after intervention
  This outcome measure will be assessed by way of surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Kuzel, MD, Principal Investigator — Virginia Commonwealth University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldberg DG, Owens-Jasey C, Haghighat S, Kavalloor S. Implementation strategies for large scale quality improvement initiatives in primary care settings: a qualitative assessment. BMC Prim Care. 2023 Nov 17;24(1):242. doi: 10.1186/s12875-023-02200-8. PMID 37978433
- See also: Quality improvement Guide — http://www.ahrq.gov/professionals/prevention-chronic-care/improve/capacity-building/pcmhqi2.html
- See also: Primary Care Facilitation Guide — https://pcmh.ahrq.gov/sites/default/files/attachments/Developing_and_Running_a_Primary_Care_Practice_Facilitation_Program.pdf
- See also: Vital Signs: Avoidable Deaths from Heart Disease, Stroke, and Hypertensive Disease - United States, 2001-2010 — http://www.cdc.gov/mmwr/preview/mmwrhtml/mm6235a4.htm?s_cid=mm6235a4_w